CLINICAL TRIAL: NCT06326762
Title: Gap CO2 in Septic Patient to Predict Cardiomyopathy Septic
Status: Completed | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Younes Oujidi, doctor, Mohammed VI University Hospital
Other Study IDs: younes
Record Dates: First submitted 2024-03-03; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Gap co2; Cardiac Output, Low; Cardiac Defect
Keywords: cardiac; CO2; septic
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myocardial Dysfunction
  Interventions: Other: comparaison
- No Myocardial Dysfunction
  Interventions: Other: comparaison

INTERVENTIONS:
Other: comparaison — description indicate

SUMMARY:
the investigators included 98 patients admitted for sepsis and septic shock (68.4% men, 31.6% women) with an average age of 60.42 years ± 15.13, ranging from 21 to 96 years. The average length of hospital stay was 7.53 days. The most noted medical histories were diabetes (38.8%), hypertension (28.6%), and renal insufficiency (17.1%). Regarding laboratory findings: the mean white blood cell count was 15,985.16 cells/mm³, the mean C-reactive protein (CRP) level was 227.69 mg/L, and the mean procalcitonin level was 50.43 µg/L. In terms of blood gas analysis: the mean lactate level was 3.67 mmol/L, and the mean PCO2 gap (DELTAPCO2) was 4.85. All our patients were continuously monitored by pulse wave analysis: the mean cardiac output was 5.69 L/min, and the mean cardiac index was 4.14 L/s/m² All our patients underwent an echocardiogram, which is a routine examination in our department and is performed at the patient's bedside. The average left ventricular ejection fraction (LVEF) was 51.73%, and the average subaortic peak velocity (ITV) was 14.66 cm.

Subsequently. the investigators examined the clinical and paraclinical profile of patients with septic cardiomyopathy. the investigators identified 19 patients with this condition, while 79 patients did not exhibit cardiac involvement. The percentage was significantly higher in the population with cardiac involvement, accounting for 28.3%. Among the patients with cardiac involvement, 76.5% had a PCO2 gap (DELTAPCO2) ≥ 6 mmHg, a significantly reduced cardiac output with an average of 3.3 L/min, and a predominantly low cardiac index, with 64.3% having an index < 2.2 L/min/m². The mortality rate was significantly increased at 73.7%.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit
* sepsis or septic shock
* at least one echocardiogram and were monitored by pulse wave contour analysis
* stay of 72 hours in the intensive care unit

Exclusion Criteria:

* Patients without sepsis or septic shock.
* Patients with COVID-19.
* Patients who died within 48 hours of hospitalization.
* Cases with incomplete medical records or patients not monitored.
* Patient with pre-existing cardiac conditions.
* post-operative patients from cardiac and thoracic surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: We included patients diagnosed with sepsis/septic shock admitted at various points in time to the intensive care units of the Mohammed VI University Hospital in Oujda.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
gapCO2 | 10 mounths
  significative in cardiomyopathy septic

CONTACTS AND LOCATIONS:
Locations (1):
- younes Oujidi, Berkane, Morocco

IPD SHARING:
Plan to Share IPD: Undecided